CLINICAL TRIAL: NCT06459986
Title: The Duration of Spinal Anaesthesia - a Prospective Observational Cohort Study
Brief Title: The Duration of Spinal Anaesthesia - a Prospective, Observational Cohort Study
Acronym: Spinalrocks
Status: Recruiting | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Aleris Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: p-2024-15423
Record Dates: First submitted 2024-06-04; First posted 2024-06-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Orthopedic Disorder
Keywords: Regional anaesthesia; Spinal anaesthesia
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal anaesthesia: Participants scheduled for orthopaedic surgery performed in spinal anaesthesia with or without sedation

SUMMARY:
Today, surgery in an ambulatory setting is preferred for many reasons. Total hip and knee arthroplasty (THA and TKA) are now procedures where patients can be sent home on the same day of the surgical procedure. However, this requires substantial knowledge of factors affecting the length of hospital stay. In this prospective, observational cohort study, we will investigate factors that affect the duration of spinal anaesthesia which is often used in THA and TKA. The aim is to gather enough data to be able to determine how local anaesthetic volume and dose affect the duration of spinal anaesthesia. This will enable us to decide whether spinal anaesthesia is a good option when performing TKA and THA in an ambulatory setting.

DETAILED DESCRIPTION:
With the increasing health care cost and the scarcity of nursing staff, there is considerable focus on providing surgery in an ambulatory setting. Total hip and knee arthroplasty (THA and TKA) are now procedures where selected patients are sent home on the same day after the procedure. Therefore, knowledge of key factors affecting the length of stay is important. One factor is the method of anaesthesia used for the operative procedure.

Spinal anaesthesia is often used for THA and TKA and has several advantages compared to general anaesthesia. However, spinal anaesthesia also has drawbacks, because it reduces the force in the legs, hindering early mobilisation. There are no good data on the duration of spinal anaesthesia. Compared to the past, there has been a shift towards using lower doses of local anaesthetic (LA) injected into the subarachnoid space. Theoretically, this should result in a shorter duration of anaesthesia, and this would be of value in an ambulatory setting. However, if the variation in the duration is high and therefore not predictable for the individual patient, spinal anaesthesia has limitations in the ambulatory setting.

The objective of the present study is to prospectively collect data on the type and dose of LA injected into the subarachnoid space and the duration of spinal anaesthesia in participants scheduled for orthopaedic surgery in spinal anaesthesia. We hypothesise that the mean duration of spinal anaesthesia is positively correlated to the dose of LA injected into the subarachnoid space.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective orthopaedic surgical procedures performed in spinal anaesthesia
* ASA 1-4.

Exclusion Criteria:

* Age < 18 years
* Anticoagulant medication therapy not paused according ESAIC/ESRA 2022 guidelines
* Local infection at the lumbar puncture site
* Bleeding disorder
* Unable to cooperate with the spinal anaesthesia procedure.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult participants scheduled for elective surgical procedures performed in spinal anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Duration of spinal anasthesia 1 | 12 hours
  Time from subarachnoid LA administration to Bromage score < 3
Duration of spinal anaesthesia 2 | 12 hours
  Time from subarachnoid LA administration to Bromage score = 1

CONTACTS AND LOCATIONS:
Overall Officials: Kai HW Lange, MD, Principal Investigator — Dept. of Anaesthesiology, Nordsjællands Hospital Hillerød, Denmark
Locations (2):
- Denmark (2):
  - Anæstesiologisk Afd, Hillerød
  - Aleris-Ringsted, Ringsted

IPD SHARING:
Plan to Share IPD: No